CLINICAL TRIAL: NCT02696694
Title: Impact of Serum Progesterone Levels on the Day of Embryo Transfer on the Success Rate in Egg Donation Cycles Under Hormonal Replacement
Brief Title: Predictive Value of Mid-luteal Serum Progesterone Levels in Egg Donation Cycles
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Elena Labarta, Elena Labarta, MD, PhD, Instituto Valenciano de Infertilidad, IVI VALENCIA
Other Study IDs: 1511-VLC-061-EL; IVI-EST-2015-01 (Other: CAEPO)
Record Dates: First submitted 2016-02-16; First posted 2016-03-02 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- P25-P75: serum progesterone between 25 and 75 percentile
  Interventions: Other: Progesterone 25-75
- <P25 ó >P75: serum progesterone <25 or >75 percentile
  Interventions: Other: Progesterone <25, >75

INTERVENTIONS:
Other: Progesterone 25-75 — Impact of serum progesterone concentrations [25-75] on the day of embryo transfer in egg donation cycles under hormonal replacement therapy
  Groups: P25-P75
Other: Progesterone <25, >75 — Impact of serum progesterone concentrations (<25, >75) on the day of embryo transfer in egg donation cycles under hormonal replacement therapy
  Groups: <P25 ó >P75

SUMMARY:
This study aims to investigate the impact of serum progesterone concentrations on the day of embryo transfer in egg donation cycles under hormonal replacement therapy. As secondary outcomes, the investigators will investigate if endometrial volume measured by three-dimensional (3D) ultrasound on the day of embryo transfer is related with progesterone levels and with chances of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age<50 yo
* BMI < 30Kg/m2
* Hormonal replacement cycle
* Endometrial thickness >6.5 mm during proliferative phase
* Transfer of one or two blastocyst grade A-B according to ASEBIR

Exclusion Criteria:

* Uterine pathology
* Cryptozoospermia
* Severe implantation failure (>6 GQ embryos transferred without success)

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients undergoing their first or second egg donation cycle
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
mid-luteal serum progesterone level | one year

SECONDARY OUTCOMES:
endometrial volume | one year

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Labarta E, Mariani G, Holtmann N, Celada P, Remohi J, Bosch E. Low serum progesterone on the day of embryo transfer is associated with a diminished ongoing pregnancy rate in oocyte donation cycles after artificial endometrial preparation: a prospective study. Hum Reprod. 2017 Dec 1;32(12):2437-2442. doi: 10.1093/humrep/dex316. PMID 29040638